CLINICAL TRIAL: NCT00225251
Title: Double-Blind Treatment of Outpatients With Dysthymic Disorder With Wellbutrin XL
Brief Title: Wellbutrin XL for Dysthymic Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St. Luke's-Roosevelt Hospital Center (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: gsk 102149
Record Dates: First submitted 2005-09-21; First posted 2005-09-23 (Estimated); Results first posted 2014-11-24 (Estimated); Last update posted 2015-11-26 (Estimated); Status verified 2014-10

CONDITIONS: Dysthymic Disorder
Keywords: Dysthymic Disorder; Dysthymia; Depression; Chronic Depression; Wellbutrin XL
MeSH Terms: conditions — Dysthymic Disorder; Depression | interventions — Bupropion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- bupropion XL (Experimental): Treatment with active medication (bupropion XL) dose ranging from 150 to 450 mg/day
  Interventions: Drug: bupropion XL
- Placebo (Placebo Comparator): Placebo comparator, matching appearance with active medication, taken from 1 to 3 tablets per day
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: bupropion XL — Antidepressant medication
  Other Names: Wellbutrin XL
  Arms: bupropion XL
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a ten-week, double-blind study of Wellbutrin XL in outpatients with dysthymic disorder, a form of low-grade chronic depression. We hypothesize that patients taking Wellbutrin XL will show greater improvement in depression symptoms and psychosocial functioning than patients taking placebo.

DETAILED DESCRIPTION:
This is a ten-week, double-blind, placebo-controlled study designed to evaluate the tolerability, dosing and efficacy of Wellbutrin XL in outpatients who meet Diagnostic and Statistical Manual-IV criteria for early onset, primary type dysthymic disorder (low-grade chronic depression). It is hypothesized that patients taking Wellbutrin XL will show greater improvement in depression symptoms and psychosocial functioning than patients taking placebo.

ELIGIBILITY:
Inclusion Criteria:

* Male and female outpatients 18-65 years of age.
* Patients with a Diagnostic and Statistical Manual Fourth Edition (DSM-IV) diagnosis of dysthymic disorder, early onset.
* Patients will have a total score of 12 or higher on the Hamilton Depression Scale (24 items) at baseline.

Exclusion Criteria:

* Patients with a DSM-IV diagnosis of Delirium, Dementia, and Amnestic, and other Cognitive Disorders.
* Patients who are pregnant or nursing women.
* Patients with a principal diagnosis meeting DSM-IV criteria for: Major Depressive disorder, Bipolar Disorder or cyclothymia, Schizophrenia, Delusional (Paranoid) Disorders and Psychotic Disorders not elsewhere classified, Severe Borderline Personality Disorder
* Patients who have a current or prior diagnosis of Anorexia Nervosa or Bulimia
* Patients who, within the past 6 months, met DSM-IV criteria for abuse of or dependence on any drug, including alcohol.
* Patients who would pose a serious risk for suicide during the course of the study, as evidenced by one of the following:

  * Report of having a specific plan for killing themselves,
  * A score of 3 or higher on the Hamilton Depression Rating Scale item #3 as rated by the treating clinician at Week 0, (indicative of active suicidal thoughts or behaviors), or
  * A suicide attempt within the past 12 months requiring emergency room visit, medical or psychiatric hospitalization, or otherwise deemed to be life-threatening (e.g. an overdose of > 1 week's dose of medication).
* Patients with a history of recurrent Grand Mal seizures or at risk of Grand Mal seizures, and those with other medical conditions in which Wellbutrin XL would be contraindicated, including a history of head trauma.
* Use of any psychotropic medication within 1 week of starting study medication
* Use of a monoamine oxidase inhibitor (a type of antidepressant) (MAOI) within the 14 days prior to the initial dose of study medication.
* Use of fluoxetine within 28 days of the initial dose of study medication.
* Use of Zyban® or other forms of bupropion hydrochloride (i.e. Wellbutrin immediate release or Wellbutrin Sustained Release (SR)) within 2 weeks of the initial dose of medication.
* Patients who have failed to respond to adequate trials (minimum of six consecutive weeks) of two different classes of antidepressant medication (see Table 1 for definitions of an adequate trial.)
* Patients with unstable medical conditions, such as acute hyperthyroidism, uncorrected hypothyroidism, undiagnosed fever, uncontrolled angina, or any other serious medical illness, including any cardiovascular, hepatic, respiratory, hematological, endocrinologic or neurologic disease, or any clinically significant laboratory abnormality.
* Patients who have begun a course of psychotherapy within 3 months of starting the study, or who plan to terminate an ongoing psychotherapy prior to the end of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2004-11; Primary Completion 2008-05 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David J. Hellerstein, MD, Principal Investigator — St. Luke's-Roosevelt Hospital Center, and NY State Psychiatric Institute
Locations (1):
- Mood Disorders Research Program, St. Luke's-Roosevelt Hospital Center, New York, New York, United States

REFERENCES:
- [Background] Hellerstein DJ, Batchelder S, Kreditor D, Fedak M. Bupropion sustained-release for the treatment of dysthymic disorder: an open-label study. J Clin Psychopharmacol. 2001 Jun;21(3):325-9. doi: 10.1097/00004714-200106000-00012. PMID 11386496
- See also: For more information about our program or this study, click here. — http://www.DepressionNY.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bupropion XL | Placebo
Started | 11 | 7
Completed | 10 | 6
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: adults with dysthymic disorder, males and females
Groups:
- Total: Total of all reporting groups
Arm/Group | Bupropion XL | Placebo | Total
Number analyzed (Participants) | 11 | 7 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.6 (11.5) | 40.0 (10.9) | 40.3 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 11
  Male | 4 | 3 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 8 | 6 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 7 | 18

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Depression Rating Scale, 24 Items (HDRS)
Description: Widely used depression rating scale, with higher scores reflecting greater level of depression. Assesses suicidality which is a safety issue.
  This study used the 24 item version of the Hamilton Depression Rating Scale; item scores range from 0 to 4 on some items, 0 to 2 or 0 to 3 on other items; range of total score = 0 to 75, with higher score indicating worse depression Response (>50% decrease) Remission (score<=7)
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bupropion XL | Placebo
Number analyzed (Participants) | 11 | 7
units on a scale | 14.4 (6.9) | 13.3 (8.4)
Statistical Analysis 1: Comparison: Bupropion XL vs Placebo; Test type: Superiority or Other; p < .05, t-test, 2 sided; Mean Difference (Net) = 3.0

2. Secondary Outcome: Cornell Dysthymia Rating Scale (CDRS)
Description: A 24 item scale assessing symptoms of chronic depression. Scores from 0 to 96 with higher score indicating worse depression
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bupropion XL | Placebo
Number analyzed (Participants) | 11 | 7
units on a scale | 26.4 (10.8) | 24 (14)

3. Secondary Outcome: Beck Depression Inventory (BDI)
Description: 21 item patient rated assessment of depression symptoms, with item scores ranging from 0 to 3. Total BDI scores can range from 0 to 63, with higher scores indicating worse depression.
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bupropion XL | Placebo
Number analyzed (Participants) | 11 | 7
units on a scale | 8 (4.4) | 12.3 (10.1)

4. Secondary Outcome: Clinical Global Improvement (CGI)
Description: A global assessment of patient improvement, ranging from 1 (very much improved) to 7 (very much worse)
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bupropion XL | Placebo
Number analyzed (Participants) | 11 | 7
units on a scale | 2.8 (1) | 2.43 (1)

5. Secondary Outcome: Global Assessment of Functioning Scale (GAFS)
Description: A clinician rated assessment of patient's overall functioning, ranging from 0 (severely impaired) to 100 (excellent functioning)
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bupropion XL | Placebo
Number analyzed (Participants) | 11 | 7
units on a scale | 64 (8.6) | 67 (9.6)

ADVERSE EVENTS:
Time Frame: 10 weeks
Description: patients were assessed for side effects over the course of the efficacy study
Arm/Group | Bupropion XL | Placebo
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/7
Other Adverse Events (participants affected / at risk) | 6/11 | 3/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bupropion XL (N=11) | Placebo (N=7)
headache (Nervous system disorders) | 4 (4) | 0 (0) — patient reported headache
dry mouth (Gastrointestinal disorders) | 3 (3) | 0 (0) — patient reported dry mouth
dizziness (Nervous system disorders) | 2 (2) | 0 (0) — patient reported dizziness
insomnia (Nervous system disorders) | 1 (1) | 3 (3) — reported difficulty sleeping

LIMITATIONS AND CAVEATS:
Early termination led to small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No